CLINICAL TRIAL: NCT02749474
Title: Maternal Cancer Diagnosis and Treatment During Pregnancy:a Registry for Maternal, Fetal, and Neonatal Outcomes With Longitudinal Follow up of Child Development and Maternal Psychological Well Being
Brief Title: Maternal Cancer Diagnosis and Treatment During Pregnancy:a Database for Maternal, Fetal, and Neonatal Outcomes
Acronym: CANCRPREGREG
Status: Recruiting | Type: Observational
Sponsor: The Cooper Health System (Other)
Responsible Party: Principal Investigator, Elyce Cardonick, Associate Dean for Research, The Cooper Health System
Other Study IDs: Cooper 15-028
Record Dates: First submitted 2016-04-13; First posted 2016-04-25 (Estimated); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Pregnancy, Cancer, Cancer in Pregnancy, Gestational Breast Cancer, Pregnancy Related
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women diagnosed with cancer: Any pregnant woman diagnosed with any cancer within 6 weeks prior to their last menstrual period, or up to 6 months after the end of their pregnancy can be enrolled.

SUMMARY:
The objective of this study is to follow the treatment options offered to pregnant women diagnosed with cancer and study the impact that their treatment or delay of treatment has on their own health and that of their children.

DETAILED DESCRIPTION:
Approximately 1:1000 pregnancies are complicated by cancer. Breast cancer is the most common type diagnosed during pregnancy. Termination of pregnancy has not demonstrated an improvement in survival. Results of an international collaborative study reported similar overall survival for patients diagnosed with breast cancer in pregnancy compared to non-pregnant patients. The consensus medical opinion supports the option to start treatment with continuation of the pregnancy. The purpose of this Cancer and Pregnancy Registry study is to prospectively follow the women diagnosed with cancer during pregnancy-collecting information about the method of diagnosis, treatment options and maternal and neonatal outcomes at delivery and yearly at follow up during childhood and adult development. Some children in this cohort have been followed up to 28 years of age.

The majority of fetal organ development is completed by 12 weeks of pregnancy, consistent with the literature showing no increased malformation rate for chemotherapy use after the first trimester of pregnancy. The central nervous system continues to develop throughout gestation and after birth. Whether chemotherapy given after the first trimester affects central nervous system maturity and results in developmental delays requires further study. The first authors to provide detailed follow up on children exposed to chemotherapy in utero were Aviles and Niz in 1988. At that time 17 children ranging in age from 4-22 years born to mothers with acute leukemia who received chemotherapy during pregnancy were examined for physical health, growth and development. Each child demonstrated normal growth and development, school performance, intelligence testing, neurological examination, and hematologic evaluation including bone marrow biopsies. This study was expanded twice. First in 1991, to 43 children ranging in age from 3 to 19 years, also after exposure in utero to chemotherapy for maternal hematologic malignancies. All children were normal physically and neurologically. School performances and standardized intelligence testing were not significantly different from controls (unrelated matched children and unexposed siblings). The same authors expanded their study again to a final report of 84 children in 2001, confirming their previous reports that chemotherapy at full doses for an aggressive hematological malignancy can be safely administered. Standardized testing on children exposed to chemotherapy was not repeated for 11 years. Drs. Amant, et al reported developmental outcomes of 70 children in Europe exposed to cancer treatment in utero. The children with developmental delays were concentrated in the group delivered preterm. In this study there was not a control group of unexposed children.

Cardonick also performed developmental testing on 57 children of women diagnosed with cancer during pregnancy, 35 were exposed to chemotherapy. Ninety-five percent of children scored within normal limits on cognitive assessments; 71% and 79% of children demonstrated at or above age equivalency in mathematics and reading scores respectively. Together Dr Cardonick and Dr Amant have evaluated children up to age 9 who were exposed to chemotherapy before birth. Reassuringly chemotherapy did not impact neurologic development, or heart performance up to age 9 years. A current study is looking at children at age 12. Studies are looking at children after exposure to both chemotherapy or radiation or cancer surgery during pregnancy. Currently Dr Cardonick is in contact with young adults in the study who are at least 18 years of age who are participating in a self-assessment tool of their physical, mental and social health. Such long follow up is what helps newly diagnosed pregnant women make informed decisions about cancer treatment during pregnancy.

Women diagnosed with cancer of any type during pregnancy can enroll voluntarily in the Cancer and Pregnancy Registry. Signed medical release forms allow the investigator to review cancer diagnostic studies and treatment course. Records are requested yearly from the treating pediatrician to follow the growth and development of the child. Participants do not have to collect their own records. All information is kept confidential. Oncologic follow up on the women is also requested yearly.

ELIGIBILITY:
Inclusion Criteria:

* Any pregnant woman diagnosed with cancer within 6 weeks before her last menstrual period or 6 months after her end of pregnancy either by delivery or miscarriage.

Exclusion Criteria:

* Women diagnosed with cancer more than 6 months after the end of a pregnancy.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cohort of pregnant women diagnosed with any type of cancer.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2003-07 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Neonatal Developmental Quotient | Yearly from 3 months to 12 years of age
  Pediatrician asked to assess developmental age compared to chronological age, ie developmental quotient

SECONDARY OUTCOMES:
Congenital Malformations | From birth to 5 years of age
  Incidence of children in registry diagnosed with birth defects after a pregnancy complicated by a cancer diagnosis.

OTHER OUTCOMES:
Mass Liquid Chromotography will be used to measure intact Taxane, Adriamycin and Cyclophosphamide chemotherapy andthe corresponding metabolites in neonatal meconium by mass liquid chromatography. | One to three specimens collected on day one of life.
  On day one of life patients who received chemotherapy during pregnancy for breast cancer can collect and submit up to 3 meconium specimens from their newborn and return in provided self addressed package with ice and all supplies provided.
Child's height percentage for age at yearly pediatric visit | Yearly until 18 years of age.
  Pediatrician surveyed yearly for child's height percentage for current age based on population normals.
Child's weight percentage for age at yearly pediatric visit | Yearly until 18 years of age.
  Pediatrician surveyed yearly for child's weight percentage for current age based on population normals.
Maternal Survival | Yearly after end of pregnancy up to 10 years.
  Oncologist surveyed yearly for maternal cancer free and overall survival
Developmental performance up to 3 years of age | 18 months of age to 3 years
  Score on Bayley Scales of Infant Development - Second Edition (BSID-III)
Developmental performance 4-7 years of age | Once when child is available between ages 4 to 7
  The Wechsler Preschool and Primary Scale of Intelligence-Revised (WPPSI-R)
Developmental performance 8 years of age and above | Once when child is available after age 8
  The Wechsler Intelligence Scale for Children, Third Edition (WISC III)
Behavioral Development at ages 1.5-5 years, 6-12 years, 17+ years | Three times during the child's life according to ages listed above.
  Parents complete the Complete Behavioral Checklist according to child's age. At age 17+ the young adult completes it themselves.
Incidence of medical conditions in children of women with cancer during pregnancy. | Yearly until 18 years of age.
  Pediatricians are asked to report any medical conditions the child is being treated for.

CONTACTS AND LOCATIONS:
Overall Officials: Elyce H Cardonick, MD, Principal Investigator — Cooper Health System
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cardonick E. Pregnancy-associated breast cancer: optimal treatment options. Int J Womens Health. 2014 Nov 4;6:935-43. doi: 10.2147/IJWH.S52381. eCollection 2014. PMID 25395871
- [Background] Cardonick E. Treatment of maternal cancer and fetal development. Lancet Oncol. 2012 Mar;13(3):218-20. doi: 10.1016/S1470-2045(11)70408-9. Epub 2012 Feb 10. No abstract available. PMID 22326923
- [Background] Cardonick E. Cancer occurs in approximately 1 per 1,000 pregnancies. Oncology (Williston Park). 2008 Jul;22(8 Suppl Nurse Ed):22-3. No abstract available. PMID 19856567
- [Background] Cardonick E, Iacobucci A. Use of chemotherapy during human pregnancy. Lancet Oncol. 2004 May;5(5):283-91. doi: 10.1016/S1470-2045(04)01466-4. PMID 15120665
- [Background] Levy C, Pereira L, Dardarian T, Cardonick E. Solid pseudopapillary pancreatic tumor in pregnancy. A case report. J Reprod Med. 2004 Jan;49(1):61-4. PMID 14976799
- [Background] Berghella V, Broth RE, Chapman AE, Cardonick E. Metastatic unknown primary tumor presenting in pregnancy as multiple cerebral infarcts. Obstet Gynecol. 2003 May;101(5 Pt 2):1060-2. doi: 10.1016/s0029-7844(02)02333-5. PMID 12738101
- [Background] Partridge AH, Pagani O, Abulkhair O, Aebi S, Amant F, Azim HA Jr, Costa A, Delaloge S, Freilich G, Gentilini OD, Harbeck N, Kelly CM, Loibl S, Meirow D, Peccatori F, Kaufmann B, Cardoso F. First international consensus guidelines for breast cancer in young women (BCY1). Breast. 2014 Jun;23(3):209-20. doi: 10.1016/j.breast.2014.03.011. Epub 2014 Apr 24. PMID 24767882
- [Background] Vandenbroucke T, Amant F. Development of children born to mothers with cancer during pregnancy: comparing in utero chemotherapy-exposed children with nonexposed controls. Am J Obstet Gynecol. 2015 Jun;212(6):830-1. doi: 10.1016/j.ajog.2015.01.035. Epub 2015 Jan 28. No abstract available. PMID 25637847
- [Background] Amant F, Vandenbroucke T, Verheecke M, Fumagalli M, Halaska MJ, Boere I, Han S, Gziri MM, Peccatori F, Rob L, Lok C, Witteveen P, Voigt JU, Naulaers G, Vallaeys L, Van den Heuvel F, Lagae L, Mertens L, Claes L, Van Calsteren K; International Network on Cancer, Infertility, and Pregnancy (INCIP). Pediatric Outcome after Maternal Cancer Diagnosed during Pregnancy. N Engl J Med. 2015 Nov 5;373(19):1824-34. doi: 10.1056/NEJMoa1508913. Epub 2015 Sep 28. PMID 26415085
- [Background] Aviles A, Diaz-Maqueo JC, Talavera A, Guzman R, Garcia EL. Growth and development of children of mothers treated with chemotherapy during pregnancy: current status of 43 children. Am J Hematol. 1991 Apr;36(4):243-8. doi: 10.1002/ajh.2830360404. PMID 1707227
- [Background] Aviles A, Neri N. Hematological malignancies and pregnancy: a final report of 84 children who received chemotherapy in utero. Clin Lymphoma. 2001 Dec;2(3):173-7. doi: 10.3816/clm.2001.n.023. PMID 11779294
- [Background] Aviles A, Niz J. Long-term follow-up of children born to mothers with acute leukemia during pregnancy. Med Pediatr Oncol. 1988;16(1):3-6. doi: 10.1002/mpo.2950160102. PMID 3340063
- [Background] Stopenski S, Aslam A, Zhang X, Cardonick E. After Chemotherapy Treatment for Maternal Cancer During Pregnancy, Is Breastfeeding Possible? Breastfeed Med. 2017 Mar;12:91-97. doi: 10.1089/bfm.2016.0166. Epub 2017 Feb 7. PMID 28170295
- [Background] Han SN, Amant F, Cardonick EH, Loibl S, Peccatori FA, Gheysens O, Sangalli CA, Nekljudova V, Steffensen KD, Mhallem Gziri M, Schroder CP, Lok CAR, Verest A, Neven P, Smeets A, Pruneri G, Cremonesi M, Gentilini O; International Network on Cancer, Infertility and Pregnancy. Axillary staging for breast cancer during pregnancy: feasibility and safety of sentinel lymph node biopsy. Breast Cancer Res Treat. 2018 Apr;168(2):551-557. doi: 10.1007/s10549-017-4611-z. Epub 2017 Dec 12. PMID 29235045
- [Background] de Haan J, Verheecke M, Van Calsteren K, Van Calster B, Shmakov RG, Mhallem Gziri M, Halaska MJ, Fruscio R, Lok CAR, Boere IA, Zola P, Ottevanger PB, de Groot CJM, Peccatori FA, Dahl Steffensen K, Cardonick EH, Polushkina E, Rob L, Ceppi L, Sukhikh GT, Han SN, Amant F; International Network on Cancer and Infertility Pregnancy (INCIP). Oncological management and obstetric and neonatal outcomes for women diagnosed with cancer during pregnancy: a 20-year international cohort study of 1170 patients. Lancet Oncol. 2018 Mar;19(3):337-346. doi: 10.1016/S1470-2045(18)30059-7. Epub 2018 Jan 26. PMID 29395867
- [Background] Borgers JSW, Heimovaara JH, Cardonick E, Dierickx D, Lambertini M, Haanen JBAG, Amant F. Immunotherapy for cancer treatment during pregnancy. Lancet Oncol. 2021 Dec;22(12):e550-e561. doi: 10.1016/S1470-2045(21)00525-8. PMID 34856152
- [Background] Amant F, Berveiller P, Boere IA, Cardonick E, Fruscio R, Fumagalli M, Halaska MJ, Hasenburg A, Johansson ALV, Lambertini M, Lok CAR, Maggen C, Morice P, Peccatori F, Poortmans P, Van Calsteren K, Vandenbroucke T, van Gerwen M, van den Heuvel-Eibrink M, Zagouri F, Zapardiel I. Gynecologic cancers in pregnancy: guidelines based on a third international consensus meeting. Ann Oncol. 2019 Oct 1;30(10):1601-1612. doi: 10.1093/annonc/mdz228. PMID 31435648
- [Background] Wolters V, Heimovaara J, Maggen C, Cardonick E, Boere I, Lenaerts L, Amant F. Management of pregnancy in women with cancer. Int J Gynecol Cancer. 2021 Mar;31(3):314-322. doi: 10.1136/ijgc-2020-001776. PMID 33649001
- [Background] Maggen C, Wolters VERA, Cardonick E, Fumagalli M, Halaska MJ, Lok CAR, de Haan J, Van Tornout K, Van Calsteren K, Amant F; International Network on Cancer, Infertility and Pregnancy (INCIP). Pregnancy and Cancer: the INCIP Project. Curr Oncol Rep. 2020 Feb 5;22(2):17. doi: 10.1007/s11912-020-0862-7. PMID 32025953
- [Background] Loibl S, Azim HA Jr, Bachelot T, Berveiller P, Bosch A, Cardonick E, Denkert C, Halaska MJ, Hoeltzenbein M, Johansson ALV, Maggen C, Markert UR, Peccatori F, Poortmans P, Saloustros E, Saura C, Schmid P, Stamatakis E, van den Heuvel-Eibrink M, van Gerwen M, Vandecaveye V, Pentheroudakis G, Curigliano G, Amant F. ESMO Expert Consensus Statements on the management of breast cancer during pregnancy (PrBC). Ann Oncol. 2023 Oct;34(10):849-866. doi: 10.1016/j.annonc.2023.08.001. Epub 2023 Aug 10. PMID 37572987
- [Background] Farooq F, Brandt JS, Cardonick E, Polushkina E, Vose J, Ahmed S, Ramakrishnan Geethakumari P, Olszewski AJ, Yasin H, Farooq U, Hamad N, Lin Y, Maggen C, Fruscio R, Gziri MM, Steffensen KD, Amant F, Evens AM. An international real-world analysis of relapsed/refractory lymphoma occurring during pregnancy. Blood Adv. 2023 Sep 26;7(18):5480-5484. doi: 10.1182/bloodadvances.2023010090. No abstract available. PMID 37259563
- [Result] Cardonick E, Gringlas M. Reply: To PMID 25434835. Am J Obstet Gynecol. 2015 Jun;212(6):831-2. doi: 10.1016/j.ajog.2015.01.036. Epub 2015 Jan 28. No abstract available. PMID 25637846
- [Result] Cardonick EH, Gringlas MB, Hunter K, Greenspan J. Development of children born to mothers with cancer during pregnancy: comparing in utero chemotherapy-exposed children with nonexposed controls. Am J Obstet Gynecol. 2015 May;212(5):658.e1-8. doi: 10.1016/j.ajog.2014.11.032. Epub 2014 Nov 27. PMID 25434835
- [Result] Cardonick E, Gilmandyar D, Somer RA. Maternal and neonatal outcomes of dose-dense chemotherapy for breast cancer in pregnancy. Obstet Gynecol. 2012 Dec;120(6):1267-72. doi: 10.1097/aog.0b013e31826c32d9. PMID 23168749
- [Result] Cardonick E, Bhat A, Gilmandyar D, Somer R. Maternal and fetal outcomes of taxane chemotherapy in breast and ovarian cancer during pregnancy: case series and review of the literature. Ann Oncol. 2012 Dec;23(12):3016-3023. doi: 10.1093/annonc/mds170. Epub 2012 Aug 8. PMID 22875836
- [Result] Henry M, Huang LN, Sproule BJ, Cardonick EH. The psychological impact of a cancer diagnosed during pregnancy: determinants of long-term distress. Psychooncology. 2012 Apr;21(4):444-50. doi: 10.1002/pon.1926. Epub 2011 Mar 2. PMID 21370310
- [Result] Cardonick E, Dougherty R, Grana G, Gilmandyar D, Ghaffar S, Usmani A. Breast cancer during pregnancy: maternal and fetal outcomes. Cancer J. 2010 Jan-Feb;16(1):76-82. doi: 10.1097/PPO.0b013e3181ce46f9. PMID 20164696
- [Result] Cardonick E, Usmani A, Ghaffar S. Perinatal outcomes of a pregnancy complicated by cancer, including neonatal follow-up after in utero exposure to chemotherapy: results of an international registry. Am J Clin Oncol. 2010 Jun;33(3):221-8. doi: 10.1097/COC.0b013e3181a44ca9. PMID 19745695